CLINICAL TRIAL: NCT03120689
Title: Learner Satisfaction and Experience With Use of a Vaginal Field Telescopic, High-definition Telescopic Camera System During Vaginal Reconstructive Procedures: A Randomized, Controlled Trial.
Brief Title: VITOM Study: A Randomized, Controlled Trial.
Acronym: VITOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Principal Investigator, Sean Francis, Chairman of Department of Obstetrics, Gynecology & Women's Health, University of Louisville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 16.0002
Record Dates: First submitted 2016-06-22; First posted 2017-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Organ Prolapse; Prolapse of Vaginal Vault After Hysterectomy; Bulging of Vaginal Wall; Incontinence; Fistula
Keywords: VITOM; Adult learners; Medical students; Residents; Vaginal surgery; Medical education
MeSH Terms: conditions — Pelvic Organ Prolapse; Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Live Surgery with VITOM (Active Comparator): Learner will not assist during the surgery, but watch the live surgery that is projected on a screen via the VITOM camera followed by a short questionnaire.
  Interventions: Other: Live Surgery using VITOM
- Live Surgery without VITOM (Active Comparator): Learner will assist in the traditional manner without the use of the VITOM camera followed by a short questionnaire.
  Interventions: Other: Live Surgery without VITOM
- Video viewing with VITOM (Active Comparator): Learner will watch a video taped using the VITOM camera followed by a short questionnaire.
  Interventions: Other: Video viewing with VITOM
- Video viewing with standard camera (Active Comparator): Learner will watch a video taped using the standard hand-held high definition camera followed by a short questionnaire.
  Interventions: Other: Video viewing with standard handheld high-definition camera

INTERVENTIONS:
Other: Live Surgery using VITOM — The vaginal operative field will be filmed with a VITOM® camera and the image from the VITOM® camera will be projected live within the operating room, so that the operating team can reference the image during the surgery.
  Arms: Live Surgery with VITOM
Other: Live Surgery without VITOM — The vaginal operation will not be filmed and learner observation will take place in the traditional way, with them looking at the physical surgical field.
  Arms: Live Surgery without VITOM
Other: Video viewing with VITOM — They will view the 10-minute standardized video filmed with the VITOM® camera.
  Arms: Video viewing with VITOM
Other: Video viewing with standard handheld high-definition camera — They will view the 10-minute standardized video filmed with the standard, handheld high-definition camera.
  Arms: Video viewing with standard camera

SUMMARY:
This is research in which students are queried by questionnaires on their satisfaction with and experience with certain educational practices (use of a camera image projecting during a live surgery) or with pre-recorded video. As data collection only involves survey data collection and satisfaction with an educational experience, and randomization/intervention is only involving use of one type of educational method versus another .

DETAILED DESCRIPTION:
As better training in vaginal surgery is a priority of gynecologic safety and quality organizations, optimizing learner satisfaction with vaginal surgery learning experiences is of paramount importance. Our purpose was to investigate if this unique camera system may have advantages in learner satisfaction both in the operating room and in video learning settings, therefore increasing the interest of the learner pool in vaginal surgery and optimizing their experience. This study has two main, non-dependent aims:

Aim 1: The investigators aim to perform a randomized, controlled trial that compares a vaginally-mounted high-definition telescopic camera system (VITOM®) that can project live images in the operating room during vaginal surgery to traditional learner surgery observation practices, with the primary outcome of learner satisfaction as measured by validated adult learner satisfaction measures.

Aim 2: The investigators aim to investigate in a randomized, controlled trial whether learners watching videos acquired with the VITOM® camera feel the video is more learner-friendly and optimal that videos acquired with traditional, tripod-mounted standard definition cameras.

ELIGIBILITY:
Inclusion Criteria:

* Adult learners (age >=18 years)
* Residents and medical students rotating in the field of gynecology at the University of Louisville and within the group of learners who are available to observe and participate in surgeries with the Urogynecologic team at any of the study sites.

Exclusion Criteria:

* Adult learners will be excluded if they have participated in the study prior, are performing a role within the surgery that precludes their participating in one of the study arms.
* If it is deemed by the surgical team that participation of the learner in the study or filming of the surgery would compromise the quality of surgery or patient safety in any manner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Learner satisfaction | 22 months
  Comparing satisfaction scores using a visual analog scale of adult learners assigned to the (VITOM®) camera group to the leaners who will be assigned to the No VITOM group during vaginal reconstructive surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Francis, M.D., Principal Investigator — University of Louisville School of Medicine
Locations (1):
- Health Care Outpatient Center and University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hobson DTG, Meriwether KV, Gaskins JT, Uddin MN, Stewart JR, Gupta AS, Francis SL. Learner Satisfaction and Experience With a High-definition Telescopic Camera During Vaginal Procedures: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):105-111. doi: 10.1097/SPV.0000000000000748. PMID 31169562